CLINICAL TRIAL: NCT00004654
Title: Phase III Randomized, Placebo-Controlled, Crossover Study of Soy Protein Isolate for Hereditary Hemorrhagic Telangiectasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Yale University (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: 199/11799; YALESM-8191
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
Keywords: genetic diseases and dysmorphic syndromes; hematologic disorders; hereditary hemorrhagic telangiectasia; rare disease
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Genetic Diseases, Inborn; Hematologic Diseases; Rare Diseases | interventions — Soybean Proteins

INTERVENTIONS:
Drug: soy protein isolate

SUMMARY:
OBJECTIVES: I. Evaluate migraine prophylaxis with soy protein isolate in patients with hereditary hemorrhagic telangiectasia.

II. Assess whether soy protein isolate reduces the frequency and severity of epistaxis and gastrointestinal bleeding in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized study. One group of patients is treated with soy protein isolate for 12 weeks. The control group receives a placebo for 12 weeks.

Patients cross to the alternate group following a 4-week washout.

ELIGIBILITY:
* Hereditary hemorrhagic telangiectasia (HHT) with 2 of the following:
* First-degree relative with HHT
* History of recurrent epistaxis or gastrointestinal bleeding
* Three or more skin telangiectasia
* Migraine headache meeting International Headache Society criteria 3 or more times a month for more than 1 year
* No pattern of daily headaches
* No severe head trauma
* No onset of headaches after 50 years of age
* At least 1 month since migraine prophylaxis
* At least 1 month since any of the following medications: Beta blockers; Calcium channel blockers; Divalproex sodium; Tricyclic antidepressants; Selective serotonin re-uptake inhibitors
* Concurrent regular treatment for migraine and gastrointestinal hemorrhage allowed
* Creatinine no greater than 2.5 g/dL
* No allergy to soy
* No pregnant women
* No women with intent to become pregnant

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Joshua R. Korzenik, Study Chair — Yale University